CLINICAL TRIAL: NCT03148509
Title: Clinical Psychopharmacology Division Institute of Mental Health, Peking University
Brief Title: A Study of Diagnosis and Treatment of Depression Based on Biological Evidence of Dopamine Reward Pathway
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Si Tianmei, Director of Clinical Psychopharmacology Division,Institute of Mental Health, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z171100000117016
Record Dates: First submitted 2017-05-08; First posted 2017-05-11 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Diagnosis and Treatment of Depression
MeSH Terms: conditions — Disease | interventions — Risperidone; Aripiprazole; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- bupropion (Experimental): receive bupropion
  Interventions: Drug: risperidone
- risperidone (Experimental): receive risperidone
  Interventions: Drug: aripiprazole
- aripiprazole (Experimental): receive aripiprazole
  Interventions: Drug: bupropion

INTERVENTIONS:
Drug: risperidone — DA receptor-mediated drugs
  Arms: bupropion
Drug: aripiprazole — DA receptor-mediated drugs
  Arms: risperidone
Drug: bupropion — DA receptor-mediated drugs
  Arms: aripiprazole

SUMMARY:
This study will recruit depressed patients unresponsive to selective serotonin reuptake inhibitor antidepressant treatment, first-degree relatives (parents or siblings) of depressed patients, schizophrenia, Parkinson's disease with and without depression, and healthy controls. The subjects need to complete the brain positron emission tomography/magnetic resonance examination, stress assessment, genetic testing, clinical evaluation and neuropsychological tests. Using the data, this study aimed to identify the abnormalities of reward circuit of depression and its differences with other diseases, and its abnormalities in first-degree relatives of depression. The depressed patients who were ineffective in treatment with selective serotonin reuptake inhibitor antidepressants were then given combined medication with dopamine receptor-mediated drugs, including dopamine transporter inhibitor - bupropion, D2 receptor antagonist - risperidone, or D2 receptor partial agonist - aripiprazole, to examine the regulation of dopamine pathway and its relationship with the therapeutic effect. Through the above work, we will provide new evidence for integrating the biological evidence of dopamine reward pathway into the clinical practice of depression.

ELIGIBILITY:
Inclusion Criteria:

* patients unresponsive to SSRI antidepressant treatment, first-degree relatives (parents or siblings) of depressed patients, schizophrenia, Parkinson's disease with and without depression, and healthy controls

Exclusion Criteria:

* Major physical illness; other DSM-IV axis I mental illness; personality disorder, mental retardation; drug and/or alcohol dependence; pregnant or lactating women; MRI examination contraindications.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression | 8 weeks

IPD SHARING:
Plan to Share IPD: No